CLINICAL TRIAL: NCT05979467
Title: The Relationship Between Serum Endocan and ADMA Levels and Penile Doppler Ultrasonography Findings in Patients With Vasculogenic Erectile Dysfunction
Brief Title: The Relationship Between Serum Endocan and ADMA Levels and Penile Doppler Ultrasonography in Erectile Dysfunction
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Cagri Akpinar, M.D., Ankara Etlik City Hospital
Other Study IDs: E-18-23-52
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Evaluation of the Relationship Between Serum Biomarkers (Endocan and ADMA) and Penile Doppler Ultrasonography Findings of Patients With Severe Erectile Dysf
Keywords: Erectile dysfunction; Endocan; ADMA; Penile Doppler
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The gold standard diagnosis in patients admitted to the hospital with the complaint of erectile dysfunction is penile doppler ultrasonography. This procedure is an invasive procedure and can cause various complications. Therefore, in this study, we aimed to support and define the diagnosis of erectile dysfunction with some biomarkers that can be measured in blood samples. At this point, we performed penile doppler ultrasonography, which is the gold standard test, for all patients who applied with the complaint of erectile dysfunction, and compared the results of penile doppler and serum biomarkers in the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe erectile dysfunction according to International Index of Erectile Function-15 questionnaire
* Patients who have not received medical or surgical treatment before
* Patients without comorbidity and related drug use

Exclusion Criteria:

* Patients who have had previous pelvic trauma or surgery,
* Patients who have benefited from using phosphodiesterase-5 enzyme inhibitors,
* Patients with psychogenic erectile dysfunction and moderate or mild erectile dysfunction according to International Index of Erectile Function-15 questionnaire,
* Patients who have neurological disease, chronic liver disease and patients with chronic renal failure and those who used drugs that could cause erectile dysfunction

Ages: 50 Years to 70 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Because erectile dysfunction is a male-specific disease
Study Population: tertiary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the relationship between serum endocan (endothelial cell-specific molecule-1), ADMA (asymmetric dimethylarginine) values and penile Doppler ultrasonography findings in patients with severe Erectile dysfunction. | 10 days from the outpatient clinic admission

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital Bilkent, Ankara, Turkey (Türkiye)